CLINICAL TRIAL: NCT05882890
Title: Does Manuel Treatment With Craniosacral Therapy Change the Experience of Dry Mouth in People Who Suffers With Dry Mouth After Cancer in Throat Ore Mouth - a Pilot Study
Brief Title: Does Craniosacraltherapy Combined With Exercises That Focuses om Respiration and Posture in the Upper Body Have an Effect on Xerostomia and Other Late Sequelae on People Who Has Been Suffering From Cancer in Mouth and Throat?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cathrine Rahbek (Other)
Collaborators: Danish Cancer Society (Other); DLHM - Danish Society for Mouth and Throat Cancer (Unknown); Danish Network for Mouth and Throat Cancer (Unknown)
Responsible Party: Sponsor-Investigator, Cathrine Rahbek, Physio Therapist, Craniotherapist cst t, Rahbek Kraniosakralterapi
Organization: Rahbek Kraniosakralterapi (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RahbekKST-PILOT
Record Dates: First submitted 2021-10-04; First posted 2023-05-31 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Xerostomia Following Radiotherapy; Xerostomia Following in Neck or Head After Cancer Surgery; Other Late Sequelae Following Radiotherapy and Cancer Surgery in Neck or Head
Keywords: craniosacral therapy; manual fascial treatment; xerostomia; late sequelae of cancer; exercises targeting posture in upper body and respiration
MeSH Terms: conditions — Xerostomia; Respiratory Aspiration | interventions — Respiration

STUDY DESIGN:
Intervention Model Description: Pilot project - single group intervention with before-after comparisons.
Masking Description: The person who does the statistic analysis will not have participated in the treatments and will not have met the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cranoisacral Therapy Receivers (Experimental): The participants will receive 50 minutes of treatment of craniosacral therapy once a week in 5 weeks. The treatment will follow the protocol "avenue of expression" end step 2c and 2c in "Ten step protocol". Instructions in home exercises is given. Before treatment the participants fill in the questionnaire "Xerostomia questionnaire after min 3 months" - a Danish standardized questionnaire of xerostomia used in hospitals. They will fill in this questionnaire again after ending their 5 treatment sessions, and again 6 months later as a follow up. They will also take notes in a diary of any side effects experienced during the treatment period. I will take their full medical history the first time we meet, I will take notes describing my treatment after every treatment session, including notes of the effects (positive and negative) that the participant has noticed.
  Interventions: Other: Craniosacral Therapy; Other: Exercices Targeting Upper Posture and Respiration

INTERVENTIONS:
Other: Craniosacral Therapy — Manual treatment, 5 grams, on the airway system, the throat, the neck, the meninges, the cranial nerve sleeves, the visceral cranium, and the soft tissue in the mouth.
  Other Names: Manual Fascial Treatment
Other: Exercices Targeting Upper Posture and Respiration — Exercises targeting upper posture and breathing exercises. The exercises is given when the therapist has reached some anatomical milestones in the treatment protocol. For example, an exercise with diaphragmatic breathing is given after manual treatment of diaphragma.

SUMMARY:
The current study aims to assess the efficacy of manual treatment with craniosacral therapy of fascial tissue in throat, neck, cranial and mouth region, on radiation and/or surgery-induced salivary gland hypofunction and xerostomia in patients who have received surgery and/or radiation therapy because of cancer in the throat and mouth regions.

The hypothesis of this project is based on a recent clinical case treated by me: I practice as a physiotherapist and craniosacral therapist in a private clinic. The patient in question was treated with craniosarcal techniques (techniques that, in a broad sense, mobilizes the fascia, including meninges, dura, sleeves around the nerve-tissue etc.). He suffered from xerostomia and hyposaliva after neck surgery and radiation therapy four years prior to my treatment. During the second treatment of fascial release of the scar tissue and of the tissue around atlas, axis and occiput the patient strongly felt that his saliva started flowing. He received an additional 3 treatments, with fascial release techniques in neck, throat meninges and mouth regions, and three months after his last treatment the patient still reported much better production of saliva than before start of treatment. Furthermore, the patient reported significant gains in ease of speaking and eating. This project aim to assess if this was only an isolated event or if craniosacral therapy could be an evidence based method to increase saliva production and decrease xerostomia for patients after surgical and radiation therapy.

DETAILED DESCRIPTION:
The aim of my project is to examine if craniosacral therapy in chest, throat, neck, cranium and mouth can decrease xerostomia in people who suffer from this after radiation therapy and/or surgery in neck or mouth because of cancer in mouth or throat. If successful, the project will be the first step in developing a clinically relevant treatment option for the growing number of patients suffering from xerostomia after radiotherapy in the throat and mouth area. This is needed, as only sub-optimal symptomatic treatments are currently available and xerostomia has been shown to reduce the quality of life. This study is inspired by a recent Danish project. In this study, stem cell therapy showed clinically significant improvements on both patient-reported measures and measured the amount of saliva produced. The authors suggest that the results may be due to a reduction of connective tissue and increased blood flow in the areas affected by radiation therapy. The authors proceed to suggest that hyperbaric oxygen treatment or other treatments attempting to increase blood flow in the radiation-affected areas could be used in combination with stem cell treatment to achieve a synergistic effect.

The hypothesis that treatment that increases the blood flow in fibrous tissue damaged after surgery or radiation has a positive effect on the tissue and its associated physiologic functions is echoed in an article about strength and shoulder mobility after breast cancer surgery. In the Danish national guidelines for breast cancer, it is also recommended that women that receive radiation therapy for their breasts because of cancer, shall receive instruction in how to treat their radiated tissue manually. The writers of the two last sources hypothesize that manual treatment of fibrous tissue damaged after surgery and radial therapy can prevent tightness in fascia and nerve tissue and preserve a proper function and mobility in shoulder and arm. The writers of the first article claims that the good results after treatment and exercises is partly attributable to the increased blood flow in the area.

A case study with 15 participants that in average 8 years previously has been through surgery or radial treatment because af cancer and who suffered from dysphagia because of fibrous tissue and neuropathy, showed that the symptoms dysphagia, airway problems and decreased mobility in the neck would be lowered by manual fascial techniques.The effect of any xerostomia was not monitored, but the study that reveals a new way to treat some of the other sequelae fibrous tissue ind mouth and neck can cause, support my hypothesis that manual treatment of fibrous tissue caused of surgery and/or radial therapy can cause increased tissue mobility, nerve conduction, and function in the fibrous tissue.

In my project I will use the treatment protocol "Avenue of expression"and a few steps from the protocol "Ten steps protocol"which addresses the areas I expect to develop fibrous tissue after radial therapy and/or surgery in neck or head. The techniques used in these protocols is light (5 grams) manual craniosacral techniques, addressing the fascia in the airway system, the neck, the throat, the meninges and nerve sleeves in the cranium, the visceral cranium, and the soft tissue in the mouth. My rationale in this project is that manual treatment of scar tissue and tissue damaged by radiation will increase mobility and blood flow and therefore possibly increase the production of saliva and decrease the sense of xerostomia.

The manual treatment is combined with home exercises that targets posture in upper body and respiration. This for maintaining the effects of the manual treatment.

Second purpose of the project is to examine if the intervention has any effect on other well-known late sequelae after treatment of cancer in mouth and neck.

Outcome is measured by a xerostomia questionaire inspired by the one used in "efficacy of the bioextra dry mouth care system in the treatment of radiotherapy induced xerostomia by Dirix P. Etal, and by selfreporting. "

My project is the very first step into supporting my hypothesis. If the results of the treatments are promising, it is my plan to continue with further research and include a placebo group and a larger sample of participants.

ELIGIBILITY:
Inclusion Criteria:

* Have finished radiation treatment and/or surgery for oro-pharyngeal head or necḱ cancer at least two years before enrolling the project
* They shall score at least 4 on an xerostomia numeric scale where 0 is no xerostomia.

Exclusion Criteria:

* Persons who by surgery have got both their submandibular saliva glands removed.
* Persons with known intercranial aneurism.
* Persons who have got a skull fracture during the last 6 months.
* Women who are trying to get pregnant.
* Persons who have sequela after a trauma on their neck that needed hospitalization.
* People with hernia on medulla oblongata.
* I will wait to treat people until after one month after they have received any dural puncture, or after 12 weeks of pregnancy.
* If I during my journal procedure of my participant finds any signs of active disease, I will send them to their doctor and do not start my treatment before the doctors approval.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathrine T Rahbek, Cst t, Principal Investigator — Rahbek KST
Locations (2):
- Denmark (2):
  - Center for Kræft og Sundhed, Copenhagen
  - - Rahbek kraniosakralterapi -FysioDanmark Skødstrup, Skødstrup, Århus

IPD SHARING:
Plan to Share IPD: Yes
The plan is to get the results released as an research article in a peer reviewed journal. If possible, the results will be accessible for everyone who is interested. I will also share it in Danish networks for interdisciplinary colleagues, and with relevant patient associations
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: I will keep the data at my desktop for at least 10 years
Access Criteria: They will be in Danish and will not be on a website - i will translate them if you contact me on my mail address.

REFERENCES:
- [Background] Hoxbroe Michaelsen S, Gronhoj C, Hoxbroe Michaelsen J, Friborg J, von Buchwald C. Quality of life in survivors of oropharyngeal cancer: A systematic review and meta-analysis of 1366 patients. Eur J Cancer. 2017 Jun;78:91-102. doi: 10.1016/j.ejca.2017.03.006. Epub 2017 Apr 18. PMID 28431302
- [Background] Gronhoj C, Jensen DH, Vester-Glowinski P, Jensen SB, Bardow A, Oliveri RS, Fog LM, Specht L, Thomsen C, Darkner S, Jensen M, Muller V, Kiss K, Agander T, Andersen E, Fischer-Nielsen A, von Buchwald C. Safety and Efficacy of Mesenchymal Stem Cells for Radiation-Induced Xerostomia: A Randomized, Placebo-Controlled Phase 1/2 Trial (MESRIX). Int J Radiat Oncol Biol Phys. 2018 Jul 1;101(3):581-592. doi: 10.1016/j.ijrobp.2018.02.034. Epub 2018 Mar 6. PMID 29678523
- [Background] Lauridsen MC, Torsleff KR, Husted H, Erichsen C. Physiotherapy treatment of late symptoms following surgical treatment of breast cancer. Breast. 2000 Feb;9(1):45-51. doi: 10.1054/brst.1999.0087. PMID 14731584
- [Background] Dirix P, Nuyts S, Vander Poorten V, Delaere P, Van den Bogaert W. Efficacy of the BioXtra dry mouth care system in the treatment of radiotherapy-induced xerostomia. Support Care Cancer. 2007 Dec;15(12):1429-36. doi: 10.1007/s00520-006-0210-y. Epub 2007 Jan 18. PMID 17235501
- See also: National Clinical Guideline for Consequences After Surgery for Breast Cancer — https://www.fysio.dk/globalassets/documents/fafo/kliniske-retningslinjer/onkologi/nkr_brystkraeft_2015.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment is done by sharing information of the project during network events for people who have been through treatment of cancer in mouth, head and/or neck. These events have been arranged by two patient associations -"DLHM" and "Netværket for Hals og Mundhulecancer" - two groups organized under the Danish Cancer Society.
Pre-assignment Details: No pre-assigment details.
Groups:
- Craniosacraltherapy Receivers: The participants will receive 50 minutes of craniosacral therapy weekly for five weeks.The treatment will follow the protocol "avenue of expression" and step 2c and 2c in "Ten step protocol" . They will get instructions in exercises targeting the upper posture and respiration to do at home between treatments. Before treatment the participants fill in the questionnaire " Xerostomia questionnaire after 3 months" - a Danish standardized questionnaire of xerostomia used in hospitals. They will fill in this questionnaire again after ending their 5 treatment sessions, and again 6 months later as follow up. They will also fill in a diary with any side effects experienced during the treatment period. I will take their full history the first time we meet, I journal my treatment after every treatment session, and journal which effects (positive and negative) the participant has noticed.
  Craniosacral therapy: Manual treatment on the whole airway system, the throat, the neck, the meninges, the cranium, nerve sleeves, the visceral cranium, and the soft tissue in the mouth.
  Exercises - targeting the upper posture and respiration.
Period: Overall Study
Arm/Group | Craniosacraltherapy Receivers
Started | 11
Completed (Eleven participants completed the treatment, but one was excluded.) | 10
Not Completed | 1
Not completed — Exclusion was due to a score in xerostomia VASscale < 4. | 1

BASELINE CHARACTERISTICS:
Groups:
- Craniosacraltherapy Receivers: Receiving 5 treatments of craniosacraltherapy , following the protocol " avenue of expression". They are also being instructed in specific exersises
Arm/Group | Craniosacraltherapy Receivers
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] — Participants were asked about their age at baseline
  years
    Age | 65.5 [40 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 6
  Sex: Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 10
results of questionaire [Mean (Full Range); unit: units on a scale] — Baseline measures in the questionnaire included an xerostomia VAS scale ranging from 0(none) - 10 (worst)
  The remaining 14 questions were phrased "how much does [question subject] bother you:" (translated from Danish) not at all (1) - a little (2) - some (3) a lot (4) very much( 5)
  The final question(number 15) were:
  "How would you feel, if you had to live the rest of your life, with the symptoms you have now?:" enjoyable(1), very satisfied (2) neither satisfied ore unsatisfied(3), very unsatisfied(4), terrible(5) the sum of points from the 15 questions gives an overall score.
  units on a scale
    VAS scale(0=best -10=worst) | 8 [6 to 10]
    Remaining 15 questions overall sum (15 worst-75 best) | 46.4 [30 to 65]
time after cancertreatment [Mean (Full Range); unit: years] | 12.5 [2 to 24]
Type of cancertreatment [Count of Participants; unit: Participants]
  laryngeal surgery | 2
  surgery in other locations (mouth,ore throat) | 6
  radiation therapy | 9

OUTCOME MEASURES:

1. Primary Outcome: Xerostomia Questionnaire
Description: A Danish questionnaire for following up on patients who have finished their cancer treatment in head and neck on a Danish hospital. It is used at least 3 months after treatment. The participants in this study has finished their treatment for cancer at least two years from enroling this study.
  VAS xerostomia scale0-10 (10 is worst) The remaining 14 questions were phrased "how much does [question subject] bother you:" (translated from Danish) not at all (1) - a little (2) - some (3) a lot (4) very much( 5)
  The final question(number 15) were:
  "How would you feel, if you had to live the rest of your life, with the symptoms you have now?:" enjoyable(1), very satisfied (2) neither satisfied ore unsatisfied(3), very unsatisfied(4), terrible(5) the sum of points from the 15 questions gives an overall score.
Time Frame: Baseline (before start of this study intervention, but at least two years after finishing treatment of cancer)
Population: 11 participants entered the project. 1 participant was not analysed, because of to low score at the xerostomia vas-scale i baseline. The inclusioncriteria for entering the analysis phase of the project was a score at at least 4 n the xerostomia vas-scale
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Craniosacral Therapy Receivers: Please refer to baseline characteristics
Arm/Group | Craniosacral Therapy Receivers
Number analyzed (Participants) | 10
score on a scale
  VAS scale(0best -10 worst) | 8 [6 to 10]
  Remaining 15 questions overall sum (15 worst-75 best) | 46.4 [30 to 65]

2. Primary Outcome: Xerostomia Questionnaire
Description: as for outcome 1
Time Frame: At the start of the fifth and last treament (intervention of this study). .
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Groups:
- Cranoisacral Therapy Receivers: The participants will receive 50 minutes of treatment of craniosacral therapy for each week in 5 consecutive weeks. The treatment will follow the protocol "avenue of expression" and step 2c and 2c in the "Ten step protocol". They will get instructions in home exercises targeting the upper posture and respiration. Before treatment the participants fill in the questionnaire "Xerostomia questionnaire after 3 months" - a Danish standardized questionnaire of xerostomia used in hospitals. They will fill in this questionnaire again after ending their 5 treatment sessions, and again 6 months later as a follow up. They will also fill in a diary with any side effects experienced during the treatment period. I will take their full history the first time we meet. I take notes of my treatment after every treatment session, including notes on which effects (positive and negative) the participant has noticed.
  Craniosacral Therapy: Manual treatment on the airway system, the throat, the neck, the meninges, the cranial nerve sleeves, the visceral cranium, and the soft tissue in the mouth.
  Exercises targeting upper posture and respiration.
Arm/Group | Cranoisacral Therapy Receivers
Number analyzed (Participants) | 10
Score on a scale
  xerostomia VAS scale(= best-10 worst) | 6.7 [3 to 10]
  the overall sum of the 15 questions questions( 15 worst-75 best) | 50.12 [35 to 69]

3. Primary Outcome: Xerostomia Questionnaire
Description: as for outcome 1
Time Frame: 6 months post after finishing the craniosacral treatment (the intervention in this study)
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Cranoisacraltherapy Receivers: The participants will receive 50 minutes of craniosacral therapy weekly in 5 weeks.The treatment will follow the protocol "avenue of expression" and step 2c and 2c in "Ten step protocol" . They will get instructions for exercises targeting the upper posture and respiration to do at home. Before treatment the participants fill in the questionnaire " Xerostomia questionnaire after 3 months" - a danish standardized questionnaire of xerostomia used of hospitals. They will fill in this questionnaire again after ending their 5 treatment sessions, and again 6 months later as a follow up. They will also fill in a diary with any side effects experienced during the treatment period. I will take their full history the first time we meet. I journalize my treatment after every treatment session, including which effects (positive and negative) the participant has noticed.
  cranio sacral therapy: Manual treatment of 5 grams on the whole airway system, the throat, the neck, the meninges, the cranium, nerve sleeves, the visceral cranium, and the soft tissue in the mouth.
  exercises- targeting the upper posture and respiration
Arm/Group | Cranoisacraltherapy Receivers
Number analyzed (Participants) | 10
score on a scale
  xerostomia VAS scale(0 best -10 worst) | 7.2 [5 to 10]
  the overall score of the 15 questions(15 worst -75 best) | 49.6 [30 to 64]

4. Secondary Outcome: Late Sequelae at Baseline
Description: A history is taken before the first treatment, where I asked if the participant suffered from 11 other well-known late seguela in this patient group.
  I asked for:
  dry mouth obstipation lymphedema tinnitus difficulty swallowing tense/stiff neck problems with respiration stiff jaw difficulty with speaking fatigue difficulty sleeping pain
  This is noted in their patient-record. Following is the number of participants who report suffering from a particular late sequelae.
Time Frame: baseline
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Cranoisacral Therapy Receivers: The participants will receive 50 minutes of craniosacral therapy weekly in 5 weeks. The treatment will follow the protocol "avenue of expression" and step 2c and 2c in "Ten step protocol" . They will get instructions in exercises targeting the upper posture and respiration to do at home. Before treatment the participants fill in the questionnaire " Xerostomia questionnaire after 3 months" - a danish standardized questionnaire of xerostomia used of hospitals. They will fill in this questionnaire again after ending their 5 treatment sessions, and again 6 months later as a follow up. They will also fill in a diary with any side effects experienced during the treatment period. I will take their full history the first time we meet, and I journalize my treatment after every treatment session, and note which effects (positive and negative) the participant has noticed.
  Craniosacral therapy: Manual treatment of 5 grams on the whole airway system, the throat, the neck, the meninges, the cranium, nerve sleeves, the visceral cranium, and the soft tissue in the mouth.
  Exercises targeting the upper posture and respiration.
Arm/Group | Cranoisacral Therapy Receivers
Number analyzed (Participants) | 10
participants
  dry mouth | 10
  obstipation | 2
  lymphedema | 3
  tinnitus | 3
  difficulty swallowing | 7
  tense/stiff neck | 5
  problems with respiration | 6
  stiff jaw | 5
  difficulty with speaking | 3
  fatigue | 3
  difficulty sleeping | 3
  pain | 1

5. Secondary Outcome: Number of Partcipants Who Experienced a Decrease in Symptoms With Their Late Sequela the 5. Time of Treatment
Description: A history is taken before the first treatment, where I asked if the participant suffered from 11 other well-known late sequela. At the 5. and last treatment I asked then if they observed any changes in their late seguela (better or worse) - They did not report any worsening of their late sequela, but a number of participants reported some positive changes.The selfreported change in symptoms is noted in their patient record. The following is the number of participants, who observed a positive change( a decrease in symptoms) in their late sequeale.
Time Frame: The 5. and last time of treatment(intervention of this study)
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Cranoisacral Therapy Receivers: The participants will receive 50 minutes treatment of craniosacral therapy weekly in 5 weeks. The treatment will follow the protocol "avenue of expression" and step 2c and 2c in "Ten step protocol". They will get instructions in exercises targeting the upper posture and respiration to do at home. Before treatment the participants fill in the questionnaire " Xerostomia questionnaire after 3 months" - a danish standardized questionnaire of xerostomia used of hospitals. They will fulfill this questionnaire again after ending their 5 treatment sessions, and again 6 months later as a follow up. They will also fill in a diary with any side effects experienced during the treatment period. I will take their full history the first time we meet. I journalize my treatment after every treatment session, and note which effects (positive and negative) the participant has noticed.
  cranio sacral therapy: Manual treatment of 5 grams on the whole airway system, the throat, the neck, the meninges, the cranium, nerve sleeves, the visceral cranium, the soft tissue in the mouth.
  exercises- targeting the upper posture and respiration.
Arm/Group | Cranoisacral Therapy Receivers
Number analyzed (Participants) | 10
participants
  dry mouth | 2
  obstipation | 2
  lymphedema | 0
  tinnitus | 0
  difficulty swallowing | 1
  tense/stiff neck | 3
  problems with respiration | 4
  stiff jaw | 0
  difficulty with speaking | 0
  fatigue | 1
  difficulty sleeping | 2
  pain | 0

6. Secondary Outcome: Number of Partcipants Who Experienced a Decrease in Symptoms With Their Late Sequela at 6 Month Follow-up
Description: A history was taken before the first treatment, where I asked if the participant suffered from 11 other well-known late sequelae in this patient group. The 5. time and 6 months after end of treatment, I asked if they observed any differences (better or worse) with their late sequelae an noted it down in their patientrecord.. They have not reported any worsening of late sequela - the following is the number of participants who reported a possitive change (a decrease in symptomps) in their late sequela at 6 month following.
Time Frame: 6 month after finishng the craniosacral treatment( intervention of this study)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cranoisacraltherapy Receivers: The participants will receive 50 minutes treatment of craniosacral therapy weekly in 5 weeks.The treatment will follow the protocol "avenue of expression" end step 2c and 2c in "Ten step protocol" . They will get instructions in exercises targeting the upper posture and respiration to do at home. Before treatment the participants fulfill the questionnaire " Xerostomia questionnaire after 3 months" - a danish standardized questionnaire of xerostomia used of hospitals. They will fulfill this questionnaire again after ending their 5 treatment sessions, and again 6 months later as a follow up. They will also fulfill a diary with any side effects experienced during the treatment period. I will take their full history the first time we meet I journal my treatment after every treatment session, and journal which effects (positive and negative) the participant has noticed.
  cranio sacral therapy: Manual treatment of 5 grams on the whole airwaysystem, the throat, the neck, the meninges, the craniel , nerve sleeves, the visceral cranium, the soft tissue in the mouth.
  exercises- targeting the upper posture and respiration
Arm/Group | Cranoisacraltherapy Receivers
Number analyzed (Participants) | 10
Participants
  dry mouth | 0
  obstipation | 1
  lymphedema | 0
  tinnitus | 0
  difficulty swallowing | 1
  tense/stiff neck | 2
  problems with respiration | 4
  stiff jaw | 0
  difficulty with speaking | 0
  fatigue | 1
  difficulty sleeping | 0
  pain | 1

ADVERSE EVENTS:
Time Frame: 5 weeks. There has not been asked for adverse events after end of treatment and there has not been reported any (through spontaneous reports while going over the trial with all participants) at 6 months follow up.
Description: Diary, asking about adverse events at every treatment. There has not been asked for adverse events after end of treatment and there has not been reported any (through spontaneous reports while going over the trial with all participants) at 6 months follow up.
Groups:
- Cranoisacraltherapy Receivers: receivers of cranoisacral therapy and home exercises
Arm/Group | Cranoisacraltherapy Receivers
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cranoisacraltherapy Receivers (N=10)
dizziness (General disorders) | 3 (4) — dizziness
irritability (General disorders) | 1 (1) — irritability
headache (General disorders) | 1 (1)
sore neck /upper back (General disorders) | 2 (2)
cramp in the neck (General disorders) | 1 (1)
sore floor of mouth (General disorders) | 1 (1)
more dislocation of the jaw than usual (General disorders) | 1 (1)
tight jaws (General disorders) | 1 (1)
difficulty controlling the tongue (General disorders) | 1 (1)
reactions on the ears (General disorders) | 2 (2)
runny nose (General disorders) | 1 (1)
more coughing and secretion than usual (General disorders) | 1 (2)
a feeling of pressure in the chest (not angina pectoris) (General disorders) | 1 (1)
more thirst (General disorders) | 1 (2)
more hungry (Gastrointestinal disorders) | 1 (1)
stomach ache/frequent visits to the toilet (General disorders) | 2 (2)
need to pee more (General disorders) | 1 (1)
feeling bloated (General disorders) | 1 (1)
feeling tired (General disorders) | 3 (4)
cramp in the feet (General disorders) | 1 (1)
restlessness in the body (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
1 participant received intervention, but was excluded before analysis because it was discovered afterwards that this participant was never eligible for inclusion (because of low score (3) in the xerostomia vas-scale at baseline - inclusion criterium was >= 4)

While scoring the xerostomia questionnaire 6 answers have inconclusive scores (either two values, or no values at all). These cases were not included when calculating the mean.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT05882890/Prot_000.pdf
  • Informed Consent Form: Informed consent for participation (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT05882890/ICF_001.pdf
  • Informed Consent Form: Informed consent for publication (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT05882890/ICF_002.pdf